CLINICAL TRIAL: NCT02233101
Title: Oral vs. Intravenous TXA Study Proposal: TJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RUSH2233
Record Dates: First submitted 2014-06-26; First posted 2014-09-08 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Blood Loss After Primary Total Joint Arthroplasty; Need for Blood Transfusion After Total Joint Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Tranexamic Acid (Active Comparator): Patients will receive either oral or intravenous Tranexamic Acid
  Interventions: Drug: Oral Tranexamic Acid
- Intravenous Tranexamic Acid (Active Comparator): Patients will receive either oral or intravenous Tranexamic Acid
  Interventions: Drug: Intravenous Tranexamic Acid

INTERVENTIONS:
Drug: Oral Tranexamic Acid — patients will receive 1950mg of oral prior to surgery to help reduce blood loss during total joint replacement
  Other Names: TXA
  Arms: Oral Tranexamic Acid
Drug: Intravenous Tranexamic Acid — Patients will receive 1950mg of intravenous Tranexamic Acid prior to total joint arthroplasty and blood loss or need for transfusion within 24 hours post operative
  Other Names: TXA
  Arms: Intravenous Tranexamic Acid

SUMMARY:
Purpose: Examine oral and intravenous Tranexamic Acid (TXA) to determine whether or not the different routes of drug administration are equivalent in terms of post-operative reduction in hemoglobin, number of transfusions, and post-operative blood loss following TJA surgery.

Hypothesis: Oral and intravenous TXA are equivalent routes of drug administration.

DETAILED DESCRIPTION:
Purpose: Examine oral and intravenous Tranexamic Acid (TXA) to determine whether or not the different routes of drug administration are equivalent in terms of post-operative reduction in hemoglobin, number of transfusions, and post-operative blood loss following TJA surgery.

Hypothesis: Oral and intravenous TXA are equivalent routes of drug administration.

Background/Scientific review:

Total hip or knee arthroplasty is associated with the risk of moderate to significant blood loss. Techniques such as the use of antifibrinolytics or desmopressin, or normovolaemic haemodilution have been used to reduce the need for allogeneic blood transfusion. Tranexamic acid (TXA) has been used to reduce blood loss and transfusion requirement for total hip and knee arthroplasty, with good results. Approximately one-third of patients undergoing total joint replacement surgery require one to three units of blood postoperatively. Tranexamic acid is a synthetic antifibrinolytic agent that has been successfully used intravenously to control bleeding after total joint replacement. The use of TXA has been shown to significantly reduce the need for blood products during total joint replacement1-4.

There are only a few studies directly comparing outcomes following the use of intravenous tranexamic acid (IVTA) and oral tranexamic acid (OTA) in arthroplasty surgery. In the randomized study by Zohar et al5. OTA (n = 20) was associated with significant allogeneic blood sparing com- pared with controls (n = 20), but not when compared with short- and long-term IVTA regimens. A recent randomized trial comparing OTA (n = 26) with placebo (n = 20) reported significant reductions in blood drained at 24 hours, and in the fall of both Hb and Hct in the OTA group, without any significant difference in the requirement of transfusion6.

Study Design: Prospective, randomized, single-blinded study

Treatment Groups:

1. Intravenous TXA Group - 1 gram IV bolus 10 minutes prior to incision
2. Oral TXA Group - 3 tablets (1950 mg) oral 2 hours prior to incision

Demographics/Patient Specifics: Age, Sex, ASA score, Weight, Height, Estimated intra-operative blood loss, Intra-operative fluids (crystalloid, colloid), Operative time, Hospitalization days, BMI, Pre-operative PT/INR, Pre-operative PTT, Pre-operative platelet count

Outcome Measurements:

1. Post-operative reduction in Hgb - Measure pre-operative Hgb levels and post-operative days 0, 1, 2, and 3 Hgb levels. Among the studies presented, they used different time points to determine the reduction in Hgb. They either used the post-operative 12-hour Hgb, post-operative day 4 Hgb, or the lowest Hgb during the hospitalization. Because we rarely have patients stay until post-operative day 4, we will have to make our measure off a different time period. We have patients get discharged as early as post-operative day 1, so we'll probably have to use the post-operative day 1 Hgb level. We feel a Hgb level difference of >1 g/dL is clinically significant.
2. Post-operative reduction in Hematocrit - Measure pre-operative and post-operative days 0, 1, 2, and 3 Hematocrit levels
3. Number of units transfused
4. Number of patients transfused
5. Cost comparison - Cost differences resulted from differences in the blood transfusion rate, length of hospital stay, and management of complications as well as from the cost of the TXA itself
6. Complications

   1. DVT or PE
   2. Return to the OR within 30 days
   3. Re-admission within 30 days
   4. Superficial infection
   5. Deep infection
   6. Periprosthetic fracture
   7. Cerebrovascular accident or Transient ischemic attack
   8. Dislocation

Risks/Benefits

The use of Tranexamic Acid is a standard of care used everyday in both primary and revision surgeries, this includes both oral and intravenous forms of Tranexamic Acid. TXA side effects include of nausea, vomiting and/or diarrhea. Gastrointestinal upset could occur with Oral tranexamic acid.

The only risk involved is the potential for breach of confidentiality and/or privacy. Below is a description of the procedure for maintaining confidentiality. There is no direct benefit to the participants in this study.

Procedures for Maintaining Confidentiality

A breach of confidentiality and/or privacy is a risk of this study. To prevent this, all collected data will be stored electronically in password-protected files to protect patient identity and information. All information will be collected and reviewed by the research team only. Data will be maintained on a password-protected computer that will be accessible only to the study team. No patient identifiers will be maintained in the database.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for a primary TKA or cementless THA with epidural/spinal anesthesia

Exclusion Criteria:

* Allergy to TXA, acquired disturbances of color vision, refusal of blood products, pre-op use of anticoagulant therapy within five days before surgery, a history of arterial or venous thromboembolic disease (such as DVT, PE, CVA, TIA), pregnancy, breastfeeding, major comorbidities (such as severe ischemic heart disease [New York Heart Association Class III or IV], previous myocardial infarction, severe pulmonary disease, renal impairment, or hepatic failure), patients who decline to participate, any patient undergoing a revision TKA, THA or BHR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig J Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Tranexamic Acid | Intravenous Tranexamic Acid
Started | 86 | 81
Completed | 74 | 80
Not Completed | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Tranexamic Acid | Intravenous Tranexamic Acid | Total
Number analyzed (Participants) | 86 | 81 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 49 | 101
  >=65 years | 34 | 32 | 66
Age, Continuous [Mean (Full Range); unit: years] | 61 [37 to 87] | 58 [30 to 85] | 60 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 38 | 33 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 81 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required Blood Transfusion
Description: Patient hemoglobin will be measured during and after surgery for the first 24 hours to determine if a blood transfusion is indicated.
Time Frame: during or within 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | Oral Tranexamic Acid | Intravenous Tranexamic Acid
Number analyzed (Participants) | 74 | 80
participants | 4 | 2

2. Secondary Outcome: Other Complications
Description: Any other complications listed below:
  1. DVT or PE
  2. Return to the OR within 30 days
  3. Re-admission within 30 days
  4. Superficial infection
  5. Deep infection
  6. Periprosthetic fracture
  7. Cerebrovascular accident or Transient ischemic attack
  8. Dislocation
Time Frame: participants will be followed for the duration of hospital stay, an expected average of no more than 30 days
Measure: Number; unit: participants
Arm/Group | Oral Tranexamic Acid | Intravenous Tranexamic Acid
Number analyzed (Participants) | 74 | 80
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Oral Tranexamic Acid | Intravenous Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/81
Other Adverse Events (participants affected / at risk) | 0/86 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes